CLINICAL TRIAL: NCT06294925
Title: Effectiveness of Etrasimod on Disease Activity and Patient-reported Outcomes in Ulcerative Colitis - EFFECT-UC
Brief Title: A Study to Learn About the Effectiveness of Etrasimod in People With Ulcerative Colitis
Acronym: EFFECT-UC
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C5041041; EFFECT-UC (Other: Alias Study Number)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Colitis, Ulcerative
Keywords: patient related outcomes; real world data; S1P modulator; Symptomatic Remission; Corticosteroid free symptomatic remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving etrasimod for ulcerative colitis
  Interventions: Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — As provided in real world practice

SUMMARY:
The purpose of this real world non-interventional study is to learn about the effects of etrasimod as treatment for patients with moderate to severe ulcerative colitis.

Patients will be treated according to standard of care and will only be included in the study if etrasimod is the best treatment choice according to the treating physician. Additionally, patients have to be between 18 and 65 years of age and should not have taken etrasimod in the past.

All patients will be prescribed etrasimod according to standard of care. Assessments will be conducted according to standard of care with the exception of health questionnaires which will be completed by the patients online on their own device.

The study duration is 52 weeks with 28 days of safety follow-up. Patients will visit their treating physician as they would if they were not enrolled in the study. During the study duration, patients will be asked to complete health questionnaires on a regular basis either on their mobile phone, tablet or computer.

The effects of etrasimod will be analyzed for each patient comparing to their disease activity prior to the start of etrasimod.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 and <65 years of age at baseline
* Patients with confirmed diagnosis of ulcerative colitis and who are prescribed etrasimod for moderately to severely active ulcerative colitis as per the product label independently of the decision to enroll a patient in this study.
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Presence of clinical findings suggestive of Crohn's disease.
* Severe extensive colitis evidenced by:

  1. Physician judgement that the patient is likely to require hospitalization for medical or surgical intervention of any kind for UC (eg, colectomy) within 12 weeks.
  2. Current evidence of acute severe UC, fulminant colitis, or toxic megacolon 3. Patients with a stoma or planned UC surgical intervention requiring hospitalization.

     4. Prior/Concomitant Therapy:

  <!-- -->

  1. any previous exposure to etrasimod including participation in the etrasimod clinical program.
  2. any co-medication with one of the following conventional therapies: methotrexate or a thiopurine (azathioprine, mercaptopurine or tioguanine) or with any of the following advanced therapies for UC: biologics (a TNF, integrin or cytokine antagonist); JAK inhibitors (filgotinib, tofacitinib or upadacitinib) or with any other S1P receptor modulator.
* Not owning a digital device with internet connection and/or not willing to complete health questionnaires on this device or not capable of using the health questionnaire collection tool.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients can be included in this study if their physician makes a clinical decision to treat them with etrasimod, as defined by the local approved label and independent from the decision to enroll the patient in this study.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with symptomatic remission | Week 12
  Symptomatic remission was defined as stool frequency sub score (SFS)= 0 (or = 1 with a ≥ 1-point decrease from baseline) and rectal bleeding sub score (RBS) =0.. Stool frequency score and rectal bleeding score are components of the Patient-Reported Outcome-2 score derived based on components of Mayo score (PRO2): instrument designed to measure disease activity of ulcerative colitis. Total score range: stool frequency 0 to 3 and rectal bleeding 0 to 3; higher score=more severe disease.
Proportion of patients with symptomatic remission | Week 52
  Symptomatic remission was defined as stool frequency sub score (SFS)= 0 (or = 1 with a ≥ 1-point decrease from baseline) and rectal bleeding sub score (RBS) =0.. Stool frequency score and rectal bleeding score are components of the Patient-Reported Outcome-2 score derived based on components of Mayo score (PRO2): instrument designed to measure disease activity of ulcerative colitis. Total score range: stool frequency 0 to 3 and rectal bleeding 0 to 3; higher score=more severe disease.

SECONDARY OUTCOMES:
Proportion of patients with clinical response | Week 12
  Clinical response was defined as decrease of at least 20% in Patient-Reported Outcome-2 score derived based on components of Mayo score (PRO2) from baseline or achievement of symptomatic remission.
Proportion of patients with clinical response. | Week 52
  Clinical response was defined as decrease of at least 20% in Patient-Reported Outcome-2 score derived based on components of Mayo score (PRO2) from baseline or achievement of symptomatic remission.
Proportion of corticosteroid-free patients with symptomatic remission | Week 52
  Symptomatic remission was defined as stool frequency sub score (SFS)= 0 (or = 1 with a ≥ 1-point decrease from baseline) and rectal bleeding sub score (RBS) =0.. Stool frequency score and rectal bleeding score are components of the Patient-Reported Outcome-2 score derived based on components of Mayo score (PRO2): instrument designed to measure disease activity of ulcerative colitis. Total score range: stool frequency 0 to 3 and rectal bleeding 0 to 3; higher score=more severe disease. Patients have to be corticosteroid-free for at least 12 weeks prior to the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- Canada (2):
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Providence Health Care (PHC), Vancouver, British Columbia
- Germany (15):
  - Gastroenterologie OpernstraBe, Kassel, Hesse
  - MVZ Gastroenterologie Aachen, Aachen
  - Praxis Heil und Müller, Andernach
  - MVZ für Gastroenterologie am Bayerischen Platz, Berlin
  - Evangelisches Krankenhaus Kalk, Cologne
  - MVZ Dachau, Dachau
  - Interdisziplinares Crohn Colitis Centrum, Frankfurt am Main
  - Facharztpraxis für Gastroenterologie, Grevenbroich
  - Studiengesellschaft BSF UG., Halle
  - Praxis für Gasteroenterologie, Heidelberg
  - Praxis für Gasteroenterologie Lübeck, Lübeck
  - Klinikum Lüneburg, Lüneburg
  - Internistische Praxengemeinschaft Oldenburg, Oldenburg
  - Magen-Darm-Zentrum Remscheid, Remscheid
  - CED am Rhein, Wesseling
- United Kingdom (14):
  - NHS Greater Glasgow and Clyde, Glasgow, Lanarkshire
  - Nottingham University Hospitals NHS Trust, Queens Medical Centre, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Western General Hospital, Edinburgh, Scotland
  - Northern Care Alliance NHS Foundation Trust, Greater Manchester, Crumpsall
  - Tunbridge Wells Hospital, Kent
  - Barts Health NHS Trust, The Royal London Hospital, London
  - St. Mark's Hospital, London
  - University College London Hospital, London
  - St Thomas' Hospital - Guy's & St Thomas' NHS Foundation Trust, London
  - Kings College Hospital, London
  - St George's Hospital - St George's Healthcare Nhs Trust, London
  - Imperial College Healthcare NHS, London
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Moran GW, Radford SJ, Walsh A, Battat R, McLean M, Kudela M, Binder E, Kulchytska N, Sahin B, Helwig U, Irving PM. Effectiveness of etrasimod on disease activity and patient-reported outcomes in ulcerative colitis-EFFECT-UC: a non-interventional, multinational, prospective cohort study protocol. BMJ Open. 2025 Dec 24;15(12):e106141. doi: 10.1136/bmjopen-2025-106141. PMID 41448713
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5041041